CLINICAL TRIAL: NCT00242333
Title: A Multi-Center Randomized, Double-Blind, Parallel Group, Placebo Controlled Study, Including an Additional Open Label Tiotropium Group, to Assess the Efficacy, Safety and Tolerability of 4 Doses of AD 237 Inhaled Once Daily for 28 Days in Subjects With COPD.
Brief Title: A Study to Assess the Safety and Efficacy of Different AD 237 Doses in Adults With COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sosei (Industry)
Collaborators: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P-AD237-005
Record Dates: First submitted 2005-10-19; First posted 2005-10-20 (Estimated); Last update posted 2006-05-16 (Estimated); Status verified 2006-05

CONDITIONS: COPD
Keywords: COPD; COAD; Chronic obstructive pulmonary disease; emphysema; chronic bronchitis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Bronchitis, Chronic

INTERVENTIONS:
Drug: AD 237

SUMMARY:
The purpose of this study is to investigate the efficacy, safety and tolerability of AD 237 in patients with chronic obstructive pulmonary disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with COPD, with symptoms of cough and chronic sputum production and/or dyspnea.
* Post-bronchodilator FEV1 at no more than 65% and at least 30% of the predicted normal value.
* Pre-bronchodilator FEV1/FVC ratio of less than 70%.
* Current or ex-smokers with a smoking history of at least 10 pack years.

Exclusion Criteria:

* History of asthma, atopy or allergic rhinitis.
* Other serious respiratory or other medical conditions which may interfere with the outcome of the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2005-10

PRIMARY OUTCOMES:
Pulmonary function

SECONDARY OUTCOMES:
Pulmonary function

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Tansley, MD, Study Director — Arakis Ltd
Locations (33):
- Bulgaria (9):
  - Specialized Hospital for Active Treatment Pneumophthysiatric Disease "Kudoglu", Plovdiv
  - Regional Dispensary for Pulmonary Diseases Rousse, Rousse
  - 5-th Multiprofile Hospital for Active Treatment, Sofia
  - MHAT "Alexandrovska", Sofia
  - Specialized Hospital for Active Treatment of Pulmonary Diseases "Sveta Sofia", Sofia
  - Central Clinical Base - Medical Institute - Ministry of the Interior, Sofia
  - Military Medical Academy, Sofia
  - UMHAT "Stara Zagora" EAD, Stara Zagora
  - University Hospital, Varna
- Hungary (9):
  - Tudogyintezete Nodradgardony, Balassagyarmat
  - III. district Outpatient Clinic, Budapest
  - Diagnostic Units Hungary Ltd, Budapest
  - Gyogyir XI. Kht.II. Tudogondozo Intezet, Budapest
  - Selye Janos Hospital, Komárom
  - Karolona Hospital, Mosonmagyaróvár
  - Szabolcs Szatmar Bereg Megyei Josa Andras Korhaz, Nyíregyháza
  - Fejer County Szent Gyorgy Hospital, Székesfehérvár
  - Vas County Markusovszky Hospital, Szombathely
- Poland (8):
  - Szpital Wojewodzki, Bielsko-Biala
  - 10 Wojskowy Szpital Kliniczny Z Poliklinika, Bydgoszcz
  - Samodzielny Publiczny Centralny Szpital Kliniczny SAM, Katowice
  - Specjalistyczny Osrodek Alergologiczny ALL-MED, Krakow
  - Barlicki University Hospital, Lodz
  - Szpital ZOZ, Oława
  - Wielkopolskie Centrum Chorob Pluc I Gruzlicy, Poznan
  - Specjalistyczna Przychodnia Lekarska "Medikard", Płock
- Romania (7):
  - Spitalul Clinic de Urgenta Floreasca, Bucharest
  - Spitalul de Pneumo Ftiziologie "Sf. Stefan", Bucharest
  - Spitalul Clinic "Colentina", Bucharest
  - Institutul National de Boli Infectioase, Bucharest
  - Spitalul Clinic de Boli Infectioase si Tropicale " Dr. Victor Babes ", Bucharest
  - Institutul de Pneumologie " Marius Nasta ", Bucharest
  - Spitalul Clinic de Urgenta Constanta, Constanța